CLINICAL TRIAL: NCT06997250
Title: Improving the Care People With Learning Disabilities Receive in Hospital: an Ethnographic Study Examining the Experiences of People With Learning Disabilities and the Organisation and Delivery of Their Care
Brief Title: Ethnography of Hospital Care for Adults With Learning Disabilities
Acronym: Care4Me
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other); University of West London (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: RHM MIS0083; NIHR206167 (Other Grant/Funding Number: National Institute for Health and Care Research)
Record Dates: First submitted 2025-04-25; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Learning Disability, Adult
Keywords: Learning disabilities; Hospital care; Acute care; Ward care
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults with learning disabilities, their carers and staff recruited from Hospital A: Adults with a learning disability receiving inpatient care in the hospital site during the data collection period
- Adults with learning disabilities their carers and staff recruited from Hospital B: Adults with a learning disability receiving inpatient care in the hospital site during the data collection period

SUMMARY:
This study will:

1. explore care experiences during a hospital admission from the perspectives of adults with learning disabilities (including people with profound learning disabilities) and their carers.
2. Examine how care is organised and delivered for adults with learning disabilities during a hospital admission.
3. Use the findings to co design guidance with people with learning disabilities, carers, and ward staff to improve care.

This study will follow the care of 8 adults with learning disabilities (including people with profound learning disabilities) during a hospital admission, in two hospitals in England. The researcher will use tailored communication to support people in sharing their experiences, including Talking Mats, Makaton and photos. The researcher will spend time with people with profound learning disabilities, learning how they communicate and carefully interpreting their non-verbal communications with their carers' support. The researcher will also talk to people's carers. The researcher will observe people's care, meetings about their care, talk to staff about their care, and read care notes (if the person agrees). The researcher will write this down and analyse it to learn how care could be improved.

The research team will work with people with learning disabilities, carers, and hospital staff to co design resources to improve ward care for people with learning disabilities. This will include:

1. recommendations to the NHS on adapting ward care;
2. a masterclass on ward care for participating hospitals;
3. a briefing to the NHS in England and the Care Quality Commission on improving how ward care is checked and managed; and
4. guidance and a toolkit on making co design more inclusive, including for people with profound learning disabilities.

The research team includes a person with a learning disability and a family carer, who will steer this project. The research team are working with people with learning disabilities and carers throughout our study to make sure it reflects their needs.

DETAILED DESCRIPTION:
This exploratory ethnographic study will examine the experiences of adults with learning disabilities and the organisation and delivery of their care during a hospital admission.

Objectives

1. Understand care experiences from the perspectives of adults with learning disabilities and family carers during a hospital admission, including adults with complex needs and profound learning disabilities.
2. Examine how care is organised and delivered for adults with learning disabilities during a hospital admission including how ward teams understand and respond to their needs.
3. Use the findings to co-design guidance with adults with learning disabilities, carers and ward staff to deliver initial strategies to improve support for adults with learning disabilities at the ward level during hospital admissions.

This project will use ethnography (with embedded case studies, observation, interviews, document analysis) to understand how care is experienced by adults with learning disabilities and how it is organised and delivered by ward teams during a hospital admission. Advisory groups of people with learning disabilities and carers of people with learning disabilities will also be involved in the analysis and interpretation of data.

The researcher will recruit 8 case studies of adults with learning disabilities (4 per hospital) who are admitted within two large general hospitals in England over a four-month period and their carers and hospital staff supporting and caring for them.

For each case study, ethnographic in situ interviews with adults with learning disabilities and family carers will be carried out to explore their experiences of care during their hospital admission. The researcher will use tailored methods of augmentative and adaptive communication for each participant and accessible interview tools. When working with participants with profound and multiple learning disabilities, the researcher will spend significant periods of time 'being with' each individual during their hospital admission to understand the meaning of each participant's "personalised forms of action" and through negotiating and interpreting meaning with their carer. The researcher will be guided by their carer(s)' advice on how best to spend time with and interact with the person and how they express a range of emotions (fear, pain, boredom, frustration, contentment). This will involve recording detailed 'micro-descriptions' of their body and facial movements, with interpretations discussed with their carer(s) during the admission.

At ward level, for each case study participant, the researcher will observe (where possible) the routine bedside care they receive during their admission. The researcher will carry out ethnographic in situ short interviews with ward staff attending the bedside and directly caring for participants to explore how they understand the participant's care and communication needs.

The researcher will carry out documentary examination of hospital passport and medical records to examine care across the admission and how it is recorded (if permission is granted).

The four-month period of data collection will deliver 160 hours of detailed ethnographic observations, across the two hospital sites. Observation periods will be carried out over three days/shifts a week across their admission, providing approximately 20 hours per case study. No identifiable data (individual names, ward names, hospital name) will be recorded during data collection. All notes will use pseudonyms for patients and carers, and staff role only will be used in notes.

The researcher will initially use maximum variation sampling. As the study progresses, sampling will include people with a learning disability who represent a range of factors that may influence care delivery, and where possible, socio-demographic factors:

* Severity of learning disability (mild to profound)
* Primary reason for the admission, including planned and unplanned admissions.
* People from Black, Asian and Minority Ethnic groups with a learning disability.
* Expected length of stay
* To include people attending hospital with differing levels of support, who have a full-time family or professional carer, or no or limited support.

The researcher will use translation services in NHS settings where required. Two forms of identification of potential case study patient participants will be used concurrently during recruitment periods.

1. Every weekday morning during data collection periods (except when active data collection is happening with a participant) Learning Disability Liaison Nurses at both hospitals will be asked to identify wards with potential participants (adults with a learning disability who are current inpatients) and wards with a planned admissions of an adult with a learning disability within the same week.
2. With the permission of matrons in both hospitals, the researcher will make weekly visits (except when active data collection is happening with a case study participant) to the nurses in charge of the medical and surgical wards on each site and any other wards identified by each site as having more people with learning disabilities attending. She will ask local nurses to screen their records for any patients with a learning disability currently on the ward.

The researcher will seek initial verbal consent from the ward manager to be present on the ward and to carry out data collection should consent be gained from the patient and their carer.

The researcher will provide potential participants (with their carers, if supporting) with accessible information sheets about the study developed with the advisory groups and advisory group lead and share a link to a video that outlines key information (via a private link on YouTube). There will an opportunity for people to ask questions about the study. For patients with learning disabilities who are assessed to lack capacity to consent, the researcher will seek advice from an appropriate consultee in line with the Mental Capacity Act. The personal consultee cannot also participate in the study as a carer. For all participants with a learning disability, the researcher will also use Dewing's model of process consent, which conceptualises consent as a continuous process with researchers considering whether a study participant is consenting to each decision across the course of the study. For people with learning disabilities who are also non-verbal, this will involve asking carer(s) how the person expresses dissent, fear or other negative emotions. The researcher will continually monitor assent, checking her interpretations with the participant's carer. If the participant or potential participant shows dissent to the researcher's presence, she will not proceed with the recruitment process. During data collection, if a participant shows dissent, that session's data collection will be ceased and participation will be reviewed with the participant and (if appropriate) their carer. If dissent continues into the next data collection session, the participant will be withdrawn from the study.

The researcher will seek written consent from the patient to access and take brief notes from their medical records and for the researcher to attend and take notes during staff meetings about their care. If they lack capacity to make these decisions, advice will be sought from their consultee. Patients can participate in the research without giving consent for their medical notes to be accessed by the researcher and/or for the researcher to make notes during meetings about their care. If consent is given for accessing medical records, or a consultee advises that they can be accessed, brief notes will be taken to outline the treatments and assessments undertaken.

It is possible that existing participants may move onto an End-of-life care pathway or into an Intensive Care Unit. If this happens, the researcher will review their participation with them with the support of their carer or personal consultee if relevant and withdraw them from the study at this point if they wish.

If a participant with a learning disability wishes to withdraw their data from the study, they can do so during the data collection period, but not afterwards. This will be discussed with all potential participants.

If the participant with a learning disability says they are happy for their carer(s) to be included, the researcher will provide the carer(s) with information and consent forms and discuss the study with them too. The carer will be required to give written consent to participate. If the carer does not wish to participate, the researcher will not collect any data about them, including during observations of the patient's care.

When consent has been gained for a patient to participate in the study, written consent will be sought from the ward manager or nurse in charge for the researcher to be present on the ward and observe care.

The researcher will sit near the patient participant during her observations, explain the study and seek verbal consent from staff. Staff members can cease participation at any point during the study.

Nursing staff will be approached at a time that does not interrupt care to ask for full written consent to participate. Should a staff member decline to give written consent, any data collected about or from them during that observation period will be destroyed and they will not be observed in any subsequent care observations. However it will not be possible to remove data about prior observations on different shifts.

Written consent from the ward manager will be sought for attending meeting discussions about the patient's care. The researcher will ask for verbal consent from all staff in the meeting and if any members of staff do not agree, she will not take notes of their contribution.

It is not practical to take consent from staff from other parts of the hospital as this may entail interrupting ward processes or interventions. Instead, posters giving information about observations on the ward will be prominently placed at the entrance to the room where observation of the patient is taking place. A note will be added to the patient's medical record to identify them as a participant in research, according to local standard research procedures. The researcher will carry information sheets and be available to answer questions and will take verbal consent from all staff when it does not interfere with clinical care processes or the work of the ward. An observation of a care interaction will be ceased should the staff member involved raise any concerns about being observed.

If the patient participant moves to another ward during data collection (including into an Intensive Care Unit) or moves onto an End-of-life care pathway, the researcher will explain the study to any new ward managers and seek initial verbal consent to continue the study on any new wards if the patient participant (or on advice from a consultee) wishes to continue. She will check that the patient and their carers (if relevant) are happy to continue with the study. She will then use the same recruitment and consent process for any new ward managers and staff as described above, for this new ward.

Analysis:

Data sets will be transcribed by the researcher into anonymised word documents or collected using handwriting software on a tablet and converted into Word files. All tablets are provided by University of Southampton and password protected. These word documents will be entered into NVivo for analysis. The goal of analysis will be to create a conceptual model of how care is organised, adapted, and delivered for people with learning disabilities during a hospital admission via: (1) a narrative approach to deliver a series (n=8) of detailed case studies that illuminate individual trajectories during an admission. (2) To analyse the ethnographic data (observation, in situ interviews, document analysis) an inductive process will be used, drawing on a grounded theory approach. (3) The ethnographic and case study analyses will be examined, refined, and brought together during the process of co-production to develop strategies to support hospital care.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a learning disability (over the age of 18)
* Receiving inpatient care in the hospital site during the data collection period

Exclusion Criteria:

* Children and young people with learning disabilities (under 18 years of age).
* People living with other kinds of cognitive impairment (not learning disability) e.g. head injury
* People not receiving inpatient care in the hospital sites during the recruitment period
* Patients on the end-of-life care pathway at the point of recruitment into the study
* Patients in intensive care units at the point of recruitment into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with learning disabilities who are inpatients in Hospital A or Hospital B during the data collection period.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Experiences of Hospital Care from the Perspectives of People with Learning Disabilities and their Carers | From enrolment in the study until end of admission (average admission is 6 days)
  Care experiences from the perspectives of adults with learning disabilities and their family carers during a hospital admission, including people with complex needs and profound learning disabilities
How Ward Care is Organised and Delivered for Adults with Learning Disabilitie | From enrolment in the study until end of admission (average admission is 6 days)
  How care is organised and delivered for adults with learning disabilities during a hospital admission including how ward teams understand and respond to their needs

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Hope, PhD, Principal Investigator — University of Southampton

IPD SHARING:
Plan to Share IPD: No
The ethnographic data collected during this study will be highly detailed and personal, making it unsuitable to be shared more widely due to the risk of identifying individuals. Participants will have consented to participate on grounds of anonymity being protected and have not consented for their IPD to be shared beyond the research team.

REFERENCES:
- See also: Funding award page (NIHR) — https://fundingawards.nihr.ac.uk/award/NIHR206167

DOCUMENTS (1):
  • Study Protocol (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT06997250/Prot_000.pdf